CLINICAL TRIAL: NCT04373538
Title: A Pilot Study for Improving Well-being by Improving Memory for Treatment for Sleep and Circadian Dysfunction
Brief Title: Improving Well-being by Improving Memory for Treatment for Sleep and Circadian Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Responsible Party: Principal Investigator, Allison Harvey, Professor, University of California, Berkeley
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: TranS-C and MSI
Record Dates: First submitted 2020-04-24; First posted 2020-05-04 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Sleep Disorder; Circadian Dysregulation
MeSH Terms: conditions — Sleep Wake Disorders; Chronobiology Disorders | interventions — Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Memory Support Intervention (Experimental)
  Interventions: Behavioral: Trans-C for sleep and circadian function + Memory Support

INTERVENTIONS:
Behavioral: Trans-C for sleep and circadian function + Memory Support — The Memory Support Intervention will be delivered interwoven with Trans-C. The Memory Support Intervention is designed to improve patient memory for treatment and involves a series of specific procedures that support the encoding and retrieval stages of episodic memory. The memory support strategies are proactively, strategically and intensively integrated into treatment-as-usual to support encoding. Memory support is delivered alongside each 'treatment point', defined as a main idea, principle, or experience that the treatment provider wants the patient to remember or implement as part of the treatment.

SUMMARY:
Mental illness is often chronic, severe, and difficult to treat. Though there has been significant progress towards establishing effective and efficient interventions for psychological health problems, many individuals do not gain lasting benefits from these treatments. The Memory Support Intervention (MSI) was developed utilizing existing findings from the cognitive science literature to improve treatment outcomes. In this study, the investigators aim to conduct an open trial that includes individuals 55 years and older to assess if a simplified version of the Memory Support Intervention improves sleep and circadian functioning, reduces functional impairment, and improves patient memory for treatment.

DETAILED DESCRIPTION:
Given the huge burden associated with mental illness, a major challenge ahead is to hasten progress toward developing and testing highly efficient and effective interventions for psychological health problems. Progress toward establishing evidence-based psychosocial treatments for most types of mental illness has been excellent, particularly the cognitive and behavioral treatments (CBT). However, much work remains. The effect sizes are moderate, gains may not persist, and there are patients who derive little or no benefit. Even under optimal conditions, treatment failure is too common. Hence, the challenge is to improve outcomes. Seminal progress toward meeting this challenge must include innovations that are safe, powerful, inexpensive and simple (for fast and effective dissemination).

The proposed research seeks to extend the investigators' program of research on one such innovation. With an R34 and an R01 from NIMH, the investigators have been seeking to improve outcome by improving memory for the content of therapy sessions. To achieve this goal, the investigators have developed and adapted existing findings from the education and cognitive science literatures. The resulting Memory Support Intervention (MSI) involves a series of specific procedures that support the encoding and retrieval stages of an episodic memory.

This line of research arises from several lines of evidence: (a) memory for the content of therapy sessions is poor and (b) memory impairment is modifiable. Although the outcomes will be relevant to psychosocial treatments for a broad range of problems, the focus of this proposal is one treatment for sleep and circadian dysfunction because (a) sleep problems are one of the most prevalent psychological health problems, (b) there is substantial and promising evidence for the efficacy of the transdiagnostic sleep and circadian (TranS-C), yet there is also room for improvement in outcome and (c) sleep problems are associated with memory impairment.

This pilot study will be conducted in order to collect data on individuals who are 55 years and older because memory functioning can decline over this phase of the lifespan. Sleep and circadian problems are also common.

The aim is: To conduct an open trial that includes n = 40 individuals 55 years and older to assess if the Memory Support Intervention (a) improves sleep and circadian functioning, (b) reduces functional impairment and (c) improves patient memory for treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 55 years and older
* English language fluency
* Exhibit a sleep or circadian disturbance as determined by endorsing 4 "quite a bit" or 5 "very much" (or the equivalent for reverse scored items) on one or more PROMIS-SD questions

Exclusion Criteria:

* Presence of an active and progressive mental or physical illness or neurological degenerative disease
* Night shift work >2 nights per week in the past 3 months
* Not able and willing to participate in and/or complete the assessments and participate in the treatment
* Current suicide risk sufficient to preclude treatment on an outpatient basis

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-06-25 (Actual)

PRIMARY OUTCOMES:
Patient-level outcome: Patient-Reported Outcomes Measurement Information System - Sleep Disturbance | Change from baseline to post-treatment, which is 8-10 weeks after the beginning of treatment
  Assesses perceived functional impairments related to sleep problems using a self-report questionnaire. The minimum value is 8. The maximum value is 40. Higher scores mean more sleep disturbance (worse outcome).
Sheehan Disability Scale | Change from baseline to post-treatment, which is 8-10 weeks after the beginning of treatment
  Assesses functional impairment on a scale from 0 to 30, where higher scores mean higher impairment

SECONDARY OUTCOMES:
Positive and Negative Affect Scale | Change from baseline to post-treatment, which is 8-10 weeks after the beginning of treatment
  Positive affect scores can range from 10-15, with higher scores representing higher levels of positive affect. Negative affect scores can range from 10-50, with lower scores representing lower levels of negative affect
Perceived Stress Scale | Change from baseline to post-treatment, which is 8-10 weeks after the beginning of treatment
  Individual scores on the Perceived Stress Scale can range from 0-40 with higher scores indicating higher perceived stress
Satisfaction with Life Scale | Change from baseline to post-treatment, which is 8-10 weeks after the beginning of treatment
  5-item instrument designed to measure global cognitive judgements of satisfaction with one's life. Scores can range from 5-35 with higher scores indicating higher levels of satisfaction with life.
Credibility Expectancy Questionnaire | At treatment Week 2 and at post-treatment which is 8-10 weeks after the beginning of treatment
  Measures the credibility and expectation of improvement from the treatment. Scores can range from 9- 81 with higher scores indicating higher treatment satisfaction.
Means and Variability of sleep efficiency (Daily Sleep Diary) | Change from baseline to post-treatment, which is 8-10 weeks after the beginning of treatment
  Daily Sleep Diary means and variability for sleep efficiency (total sleep time/time in bed X 100), Total sleep time (TST), Total wake time (TWT), bedtime, waketime.
Patient-Reported Outcomes Measurement Information System - Sleep Related Impairment | Change from baseline to post-treatment, which is 8-10 weeks after the beginning of treatment
  Assesses perceived functional impairments related to sleep problems in a self-report questionnaire. The minimum value is 16. The maximum value is 80. Higher scores mean more sleep related problems (worse outcome).
Composite Sleep Health Score | Change from baseline to post-treatment, which is 8-10 weeks after the beginning of treatment
  Composite Sleep Health Score which is defined as the sum of scores on 6 sleep health dimensions: Regularity (Midpoint fluctuation), Satisfaction (Sleep quality question on PROMIS-SD), Alertness (Daytime sleepiness question on PROMIS-SRI), Timing (Mean midpoint), Efficiency (Sleep efficiency) and Duration (Total Sleep Time).
British Columbia Complaints Inventory | Change from baseline to post-treatment, which is 8-10 weeks after the beginning of treatment
  Assessed perceived cognitive difficulties, scale consists of 6 items. Scores can range from 0-18 with higher scores indicating higher levels of perceived cognitive difficulties
Mutlidimensional Fatigue Inventory | Change from baseline to post-treatment, which is 8-10 weeks after the beginning of treatment
  20-item scale designed to evaluate five dimensions of fatigue. Scores can range from 20-100 with higher total scores corresponding with more acute levels of fatigue
Cognitive Failures Questionnaire | Change from baseline to post-treatment, which is 8-10 weeks after the beginning of treatment
  Used to assess the frequency with which people experienced cognitive failures. Scores range from 0-100, with higher scores indicating higher levels of cognitive failures.
Epworth Sleepiness Scale | Change from baseline to post-treatment, which is 8-10 weeks after the beginning of treatment
  Used to assess daytime sleepiness. Scores can range from 0-24 with higher scores indicating higher levels of daytime sleepiness.
Memory for Treatment | At post-treatment, which is 8-10 weeks after the beginning of treatment
  Recall on the Patient Treatment Recall Task
Generalization Task Questionnaire | Change from baseline to post-treatment, which is 8-10 weeks after the beginning of treatment
  Measures how treatment gains sustained during therapy have generalized to the participant's thinking and functioning during every day life
Acceptability Intervention Measure | Through therapy completion, an average of 8 weeks
  Assess provider perceptions of the appropriateness of the treatment intervention using a self-report questionnaire
Intervention Appropriateness Measure | Through therapy completion, an average of 8 weeks
  Assesses provider perceptions of the appropriateness of the treatment intervention using a self-report questionnaire
Feasibility of Intervention Measure | Through therapy completion, an average of 8 weeks
  Assesses provider perceptions of the feasibility of the intervention using a self-report questionnaire

OTHER OUTCOMES:
STOP-BANG Questionnaire | Baseline only
  Scores range from 0-8 with higher scores associated with higher risk of experiencing sleep apnea
Screen for periodic limb movement disorder | Baseline only
  Restless Leg Syndrome Questions
Medication Dosage | Change from baseline to post-treatment, which is 8-10 weeks after the beginning of treatment
  Collect dose, type, frequency and changes in medications
Medication Type | Change from baseline to post-treatment, which is 8-10 weeks after the beginning of treatment
Medication Use Frequency | Change from baseline to post-treatment, which is 8-10 weeks after the beginning of treatment
Change in Medications | Change from baseline to post-treatment, which is 8-10 weeks after the beginning of treatment
Semi-structured interview | Only at post-treatment which is 8-10 weeks after the beginning of treatment
  Assess patient perceptions of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Allison Harvey, PhD, Principal Investigator — University of California, Berkeley
Locations (1):
- University of California, Berkeley, Berkeley, California, United States